CLINICAL TRIAL: NCT03758079
Title: Comparison of Gabapentin With Doxepin in the Management of Uremic Pruritus: Pilot Study
Brief Title: Comparison of Gabapentin With Doxepin in the Management of Uremic Pruritus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Balamand (Other)
Responsible Party: Principal Investigator, Julien Bachour, MD, Principle Investigator, University of Balamand
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 064-17/717
Record Dates: First submitted 2018-11-19; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Uremic Pruritus
MeSH Terms: interventions — Doxepin; Gabapentin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxepin (Active Comparator): 10 mg Doxepin daily for 4 weeks
  Interventions: Drug: Doxepin
- Gabapentin (Active Comparator): Gabapentin 100mg after each dialysis session
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Doxepin — 10 mg Doxepin for 4 weeks
  Other Names: Silenor; Sinequan; Adapin
  Arms: Doxepin
Drug: Gabapentin — dose of 100mg after each hemodialysis session (increased as tolerated) for 4 weeks
  Other Names: Neurontin; Gralise; Gabarone; Fanatrex
  Arms: Gabapentin

SUMMARY:
This is a single blind randomized trial to compare efficacy and side effects of Gabapentin with Doxepin. Hemodialysis patients with uremic pruritus at one dialysis center of Saint George Hospital University Medical Centre were included in this study. Patients were divided into 2 groups to receive either 10 mg Doxepin daily or Gabapentin at a dose of 100mg after each hemodialysis session (increased as tolerated) for 4 weeks, after which patients were treated reversley. Pruritus severity and its effect on quality of life will be assessed by using visual analog scale (VAS), 5-D pruritus scale and dermatology life quality index (DLQI). Include patients will have to fill these forms at baseline and at end of week1, week2 and week4

DETAILED DESCRIPTION:
Pruritus is one of the frustrating skin manifestations of advanced renal failure. Many options have been used for the management of uremic pruritus (UP) such as Pregabalin, Gabapentin, Doxepine and Desloratidine. Gabapentin, a GABAergic drug, has been found to be effective in the treatment of uremic pruritus. Doxepin, a potent antihistamine drug, is used orally or topically in many pruritic conditions such as UP, idiopathic pruritus, atopic dermatitis, neurogenic, or psychogenic pruritus and, in the management of the UP in hemodialysis patients.

No comparative head to head study between Gabapentin and Doxepine has been conducted to date. The aim of this study was to compare Gabapentin and Doxepin in treatment of uremic pruritus in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* prevalent patients undergoing HD with UP for at least three months
* any medications with antipruritic effects to be discontinued one week before the study
* Hemodialysis performed for 3-4 h thrice weekly via a low flux polysulphonedialyser [1.3-1.6 m2 surface areas] using bicarbonate and/or acetate dialysis fluid
* well controlled Calcium, Phosphorus and iPTH levels

Exclusion Criteria:

* patients labeled high risk of fall (Having a score more than 16/20 using part 1 from Falls Risk Assessment Tool (FRAT)
* patients taking drugs that interact with doxepin or gabapentin
* patients with hepatic failure
* patients with hyperthyroidism
* patients with narrow angle glaucoma
* patients with heart block or decompensated heart failure or hypotension (defined as systolic blood pressure less than 90 mmHg) or myocardial infarction in the past three months
* history of allergy to gabapentin or doxepin
* uncontrolled psychiatric diseases
* pregnant patients
* patients with psoriasis, atopic dermatitis or any other condition that can justify the pruritus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Worst-itching Visual Analog Scale (VAS) at week 4 | 1, 2, 4 weeks
  a 10cm horizontal line marked from zero (no pruritus) to 10 (worst possible pruritus). The pruritus will be assessed subjectively and scored as follows: no pruritus (VAS score 0), mild (VAS score 1-3) with episodic and localized pruritus without disturbance in usual work and sleep, moderate (VAS score 4-7) with generalized and continuous pruritus without sleep disturbance and severe (VAS score 8-10) with generalized, continuous pruritus and sleep disturbance.
Change from baseline in 5-D Itch Scale score at week 4 | 1, 2, 4 weeks
  multidimensional questionnaire. The five dimensions are degree, duration, direction, disability and distribution. The scores of each of the five domains will be achieved separately and then summed together to obtain a total 5-D score ranging between five (no pruritus) and 25 (most severe pruritus). For the distribution domain, the number of affected body parts is tallied (potential sum 0-16) and the sum is sorted into five scoring bins: sum of 0-21⁄4score of 1, sum of 3-51⁄4score of 2, sum of 6-101⁄4score of 3, sum of 11-131⁄4score of 4 and sum of 14-161⁄4score of 5
Change from baseline in Dermatology life quality index (DLQI) at week 4 | 1, 2, 4 weeks
  10-Item questionnaire evaluating: impact of skin condition on HRQoL during the past week, symptoms and feeling, daily activities, leisure, work and school, personal relationships, treatment. A Score range from 0 to 30.

SECONDARY OUTCOMES:
side effects of each treatment | 4 weeks
  Number of patients who report side effects while on each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger N Haber, MD, Principal Investigator — University of Balamand/Saint George Hospital University Medical Center
Locations (1):
- Saint George Hospital University Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided